CLINICAL TRIAL: NCT03447743
Title: Re-entry XR-NTX for Rural Individuals With Opioid Use Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Michele Staton (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Michele Staton, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R34DA045856-01 (NIH); R34DA045856-01 (NIH)
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- XR-NTX services as usual (Other): Participants will receive on-going XR-NTX injections in a local community clinic
  Interventions: Drug: XR-NTX community location

INTERVENTIONS:
Drug: XR-NTX community location — XR-NTX will be administered at the local health care clinic
  Other Names: Vivitrol

SUMMARY:
The overall aim of this R34 proposal is to examine the feasibility, acceptability, and short-term outcomes associated with an innovative service delivery model to increase adherence to extended-release naltrexone (XR-NTX) during the transition from jail to the community for rural individuals with opioid use disorder (OUD). The significance of this study is grounded in the public health emergency associated with the opioid epidemic in rural Appalachia, the increased vulnerability of rural individuals with OUD, and the dearth of available and accessible evidence-based treatment in the region. This study has potential to make a significant contribution to the OUD treatment field by advancing knowledge on innovative service delivery models to increase access to evidence-based treatment to reduce the prevalence of opioid use disorders and related health disparities among hard-to-reach, high-risk, underserved populations.

DETAILED DESCRIPTION:
The overall aim of this R34 proposal is to examine the feasibility, acceptability, and short-term outcomes associated with an innovative service delivery model to increase adherence to extended-release naltrexone (XR-NTX) during the transition from jail to the community for rural individuals with opioid use disorder (OUD). The significance of this study is grounded in the public health emergency associated with the opioid epidemic in rural Appalachia, the increased vulnerability of rural individuals with OUD, and the dearth of available and accessible evidence-based treatment in the region. This R34 has potential to make a significant contribution to the OUD treatment field by advancing knowledge on innovative service delivery models to increase access to evidence-based treatment to reduce high-risk opioid use and related health disparities among hard-to-reach, high-risk, underserved populations. The study will be accomplished through two specific aims: (1) Adapt XR-NTX services for use in community supervision (P&P) offices to increase adherence during re-entry from jail for rural individuals with OUD. (2) A small scale pilot will be conducted to examine feasibility, acceptability, and short-term outcomes of the adapted protocol on XR-NTX adherence and relapse to opioid use. Rural justice-involved individuals on community supervision with OUD will be invited to initiate XR-NTX and continue injections for up to three months in the community. If this study establishes feasibility of this innovative community-based treatment model for XR-NTX in a rural, underserved area, findings will be used to develop an R01 application to test the approach in a larger RCT during community re-entry from jail among high-risk rural individuals with OUD in Appalachia. The long-term goal of this research is to increase access to evidence-based treatment for OUD among high-risk, underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for opioid use disorder
* Anticipated release date within 30 days
* Opioid free
* Not currently in methadone or buprenorphine trial
* No serious medical or psychiatric condition
* Willingness to enroll in the trial

Exclusion Criteria:

* Positive study pregnancy test
* Abnormal liver function tests (5X upper limits of normal)
* Chronic pain conditions that require opioid therapies
* Untreated medical or psychiatric disorder
* Suicidal ideation
* BMI > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Staton, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended Release Naltrexone (XR-NTX) Services as Usual: Participants will receive on-going XR-NTX injections in a local community clinic
  XR-NTX community location: XR-NTX will be administered at the local health care clinic
Period: Overall Study
Arm/Group | Extended Release Naltrexone (XR-NTX) Services as Usual
Started | 9
Completed | 2
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 1
Not completed — Did not meet criteria to continue | 1

BASELINE CHARACTERISTICS:
Arm/Group | Extended Release Naltrexone (XR-NTX) Services as Usual
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 36.1 [22 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Ever Been in a Substance Use Treatment Program [Count of Participants; unit: Participants] | 5
Ever Prescribed Medication for Opioid Use Disorder [Count of Participants; unit: Participants] | 4
Ever Injected any Drug [Count of Participants; unit: Participants] | 8
Ever Overdosed [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Study Enrollment
Description: Study enrollment is defined as the number of participants who initiate XR-NTX.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | XR-NTX Services as Usual
Number analyzed (Participants) | 9
Participants | 7

2. Secondary Outcome: Number of Participants With Opioid Relapse
Description: The short-term outcome of interest includes any relapse to opioid use (any use of opioids by self-report and urine drug screen; continuous measure of number of days of use).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | XR-NTX Services as Usual
Number analyzed (Participants) | 9
Participants | 3

ADVERSE EVENTS:
Time Frame: 3 months
Description: AEs were assessed by medical staff and at follow-up based on participant self-report.
Arm/Group | XR-NTX Services as Usual
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XR-NTX Services as Usual (N=9)
Hospitalization (Hepatobiliary disorders) | 1 (1) — Participant was hospitalized and received a possible cirrhosis diagnosis, which was determined to not be related to study participation. Participant was discontinued from the study.
Hospitalization (Injury, poisoning and procedural complications) | 1 (1) — Participant was hospitalized following an altercation

LIMITATIONS AND CAVEATS:
* Number of individuals re-entering the community onto supervision in the specified county
* Overall small sample size that was able to be recruited
* COVID-19 (coronavirus) shut down recruiting in criminal justice settings for part of the study period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT03447743/Prot_ICF_000.pdf